CLINICAL TRIAL: NCT03749148
Title: A Randomized, Double-blind, Placebo-controlled, Proof of Concept, Multicenter, 16-week Treatment Study With a 16 Week Follow-up Period to Assess the Efficacy and Safety of Dupilumab (Anti-IL4Ra) in Adult Patients With Cholinergic Urticaria Despite H1-antihistamine Treatment
Brief Title: Cholinergic Urticaria - Efficacy of Dupilumab
Acronym: CHED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sanofi (Industry); Proinnovera GmbH (Industry)
Responsible Party: Principal Investigator, Marcus Maurer, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-001-02; 2017-001262-25 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-11-21 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Cholinergic Urticaria
Keywords: hives; itch; exercise
MeSH Terms: conditions — Urticaria; Pruritus; Motor Activity | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Phase 2 multicenter, randomized, double blind, placebo controlled, proof of concept, parallel group, two-arm, investigator-initiated trial (IIT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Active Comparator): Dupilumab, s.c. administration 2 injections (600mg) as loading dose, 1 injection (300mg) every 14 days for a total of 16 weeks
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): matching Placebo, s.c. administration 2 injections as loading dose, 1 injection every 14 days for a total of 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — anti-IL4-Receptor alpha
  Arms: Dupilumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy in reducing disease activity and safety of Dupilumab in adult patients with cholinergic urticarial (CholU) who are symptomatic despite H1-antihistamine treatment (licensed dose).

DETAILED DESCRIPTION:
Treatment with Dupilumab has been shown to reduce clinically significant exacerbations and to improve skin symptom control as well as quality of life in moderate to severe atopic dermatitis patients and in moderate to severe asthma patients. It has been approval by European Medicines Agency (EMA) for the treatment of atopic dermatitis patients in September 2017.

Dupilumab is a novel monoclonal antibody that inhibits interleukin-4 (IL-4) and interleukin-13 (IL-13) signaling and was previously found to be effective in atopic dermatitis and asthma. Considering that CholU and atopic diseases share many common features (e.g. key pathogenic role of mast cells and immunoglobulin E (IgE), itch is a dominant symptom, Th2 dominance), it is reasonable to expect that Dupilumab is beneficial in CholU.

These results suggest that Dupilumab may provide an effective treatment option for patients with insufficient treatment responses to H1-antihistamines exhibiting wheal and flare type skin reactions.

The gold standard treatment of CholU consists of administration of antihistamines. In most patients, symptoms persist with standard dosing of antihistamines. In antihistamine-refractory patients with cholinergic urticaria, no other licensed treatment is currently available. In 2014, omalizumab has been licensed for add-on therapy in chronic spontaneous urticaria (CSU) patients who still have symptoms despite standard-dosed antihistamine treatment, but not for chronic inducible forms of urticaria. Accordingly, there is still a great medical need for additional treatment options of CholU patients that are refractory to antihistamine treatment.

Dupilumab has excellent potential to provide symptom control in CholU. This study will provide additional valuable insights into the therapeutic potential of Dupilumab in improving quality of life in these patients, in addition to managing CholU symptoms.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: cholinergic urticaria (ongoing disease)

1. Patient is informed about study procedures and medications and has given written informed consent before any assessment.
2. Patient is able to communicate with the investigator, understands and complies with the requirements of the study.
3. Male or Female
4. Patient is 18-75 years of age
5. Patient is diagnosed with CholU and refractory to standard of care treatment at the time of randomization, as defined by the following:

   The presence of itch and hives for equal or more than 6 consecutive weeks at any time prior to enrollment despite current use of licensed dose H1 antihistamine Urticaria control test UCT less than 12 prior to randomization (Day 1) CholU diagnosis for 6 months
6. Willing and able to complete a daily symptom diary for the duration of the study and adhere to the study visit schedules.
7. Patients must not have more than one missing diary entry in the 7 days prior to randomization. Re-screening may be considered.
8. Women of childbearing potential have to agree to use an acceptable form of contraception (as determined by the site investigator) and have to continue its use for the duration of the study.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
2. History of hypersensitivity to any of the study drugs (Dupilumab, rescue medication) or their components or to drugs of similar chemical classes.
3. Clearly dominating other form of urticaria as etiology for wheal and flare type reactions. This includes the following: Chronic spontaneous urticaria, inducible urticaria: urticaria factitia, cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic, or contact-urticaria. These diseases are allowed as comorbidities, if cholinergic urticaria is the dominating form of chronic urticaria.
4. Other diseases with symptoms of urticaria or angioedema, including urticaria vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema (e.g., due to C1 inhibitor deficiency)
5. Any other active skin disease associated with chronic itching that might confound the study evaluations and results (e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, etc.)
6. Patients who have received concomitant prohibited medication within the last 3 months prior to screening:

   * Anti-IgE therapy (e.g. omalizumab)
   * Routine (daily or every other day during 5 or more consecutive days) doses of systemic corticosteroids or other immunosuppressants
   * Intravenous immunoglobulins
   * Biological therapy
   * Systemic immunosuppressants
   * Live/attenuated vaccines
   * Other investigational drugs
7. Use of prohibited treatment detailed in protocol (see section 6.5.8 and Table 3: Prohibited treatment).
8. History of anaphylactic shock.
9. Presence of hypereosinophilic diseases (blood eosinophils >1500 cells/mm3 at the latest available test).
10. Presence of clinically significant cardiovascular, bronchial, neurological, psychiatric, metabolic or other pathological conditions that could interfere with the interpretation of the study results and/or compromise the safety of the patients.
11. Medical examination or laboratory findings that suggest the possibility of decompensation of co-existing conditions for the duration of the study. Any items that are cause for uncertainty must be reviewed with the Medical Monitor.
12. Inability to comply with study and follow-up procedures.
13. History of malignancy of any organ system (other than localized basal cell carcinoma or actinic keratosis or Bowen disease: carcinoma in situ of skin; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
14. Evidence of severe renal dysfunction at screening
15. Patient considered potentially unreliable or where it is envisaged the patient may not consistently attend scheduled study visits.
16. Serious psychiatric and/or psychological disturbances.
17. History or evidence of ongoing drug or alcohol abuse, within the last 6 months prior to randomization.
18. Patient unable to complete a patient diary or complete questionnaires on paper.
19. Any other condition or prior/current treatment, which in the opinion of the investigator renders the patient ineligible for the study schedule.
20. Study personnel or first degree relatives of investigator(s) must not be included in the study.
21. Subjects who live in detention on court order or on regulatory action as per local and national law (see §40 subsection 1 sentence 3 no. 4 Arzneimittelgesetz)
22. Pregnant or nursing (lactating) women, where pregnancy is defined
23. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropi (hCG) laboratory test.
24. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are using highly-effective methods of contraception during the duration of the study. Highly-effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient), Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
    * Male sterilization (at least 6 m prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS) In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum (follicle-stimulating hormone) FSH levels > 40 (milli international units) mIU/mL; or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six months ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
25. Patients with active confirmed SARS -CoV2 infection are to be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
cholinergic Urticaria activity score over 7 days (CholUAS7) | Change from 7 days prior to baseline (Visit (V) 1) to 7 days prior to week 16 (V9)]
  0-42 points total range, higher values equal more disease activity

SECONDARY OUTCOMES:
Global assessment | Change from 7 days prior to baseline (Visit (V) 1) to 7 days prior to week 16 (V9)]
  Global assessment (physician and patient) by visual analogue score (VAS; 0 - no pain; 10 - max. amount of pain) for disease activity
provocation urticaria activity score (pUAS; 0 - no activity; 3 - high activity) | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  Reduction in provocation urticaria activity score
weekly pruritus score (PS7; 0 - no activity; 21 - high activity) | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  Reduction in weekly pruritus score (PS7)
Responder rates and sypmtom patterns | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  symptoms assessed by diary
Urticaria control test, dermatological quality of life, cholinergic urticaria quality of life | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  Quality of life instruments as assessed by urticaria control test (UCT; 16 - complete disease control; 0 - max. amount of physical symptoms), dermatological quality of life (DLQI; 0 - no impairment of life quality, 30 - maximum impairment) , and cholinergic urticaria quality of life (CholUQoL; 0 - no impairment; 120 - worst impairment)
Use of rescue medication | Change from 7 days prior to baseline (V1) to 7 days prior to week 16 (V9)]
  frequency of how often rescue medication was used

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (8):
- Germany (8):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Giessen und Marburg, Marburg, Hesse
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Hautklinik Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Hautklinik der Universitätsmedizin Mainz Clinical Research Center, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein, Klinik für Dermatologie, Venerologie und Allergologie, Kiel, Schleswig-Holstein
  - Charité-Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No